CLINICAL TRIAL: NCT03538015
Title: The Use of Low-Dose Carvedilol to Improve Hypoglycemia Awareness in Patients With Type 1 Diabetes Mellitus
Brief Title: Carvedilol in Treating Hypoglycemia Unawareness
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor was impacted by COVID-19 and did not have sufficient funds to continue.
Sponsor: Owen Chan, PhD (Other)
Responsible Party: Sponsor-Investigator, Owen Chan, PhD, Associate Professor of Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #108879
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2020-09-09 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Hypoglycemia Unawareness
Keywords: Type 1 Diabetes Mellitus; β-blocker
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled study in patients with Type 1 diabetes mellitus and hypoglycemia unawareness
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Carvedilol 3.125 mg (Experimental): After enrollment, participants will be placed on continuous glucose monitoring (CGM). One week after CGM placement, participants will undergo the first hypoglycemic clamp study to obtain baseline measures of hypoglycemia frequency, hypoglycemia awareness scores and hormone responses. Following the initial clamp procedure, participants will receive 4 weeks of low-dose carvedilol treatment. After 4 weeks of treatment, the participants will undergo a second hypoglycemic clamp session.
  Interventions: Drug: Carvedilol 3.125 mg
- Carvedilol 2.5 mg (Experimental): After enrollment, participants will be placed on continuous glucose monitoring (CGM). One week after CGM placement, participants will undergo the first hypoglycemic clamp study to obtain baseline measures of hypoglycemia frequency, hypoglycemia awareness scores and hormone responses. Following the initial clamp procedure, participants will receive 4 weeks of low-dose carvedilol treatment. After 4 weeks of treatment, the participants will undergo a second hypoglycemic clamp session.
  Interventions: Drug: Carvedilol 2.5 mg
- Placebo capsule (Placebo Comparator): After enrollment, participants will be placed on continuous glucose monitoring (CGM). One week after CGM placement, participants will undergo the first hypoglycemic clamp study to obtain baseline measures of hypoglycemia frequency, hypoglycemia awareness scores and hormone responses. Following the initial clamp procedure, participants will receive 4 weeks of placebo treatment. After 4 weeks of treatment, the participants will undergo a second hypoglycemic clamp session.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Carvedilol 3.125 mg — Participants will receive a 3.125 mg oral dose of carvedilol twice daily during the 4-week treatment period
  Other Names: Coreg
  Arms: Carvedilol 3.125 mg
Drug: Carvedilol 2.5 mg — Participants will receive a 2.5 mg oral dose of carvedilol twice daily during the 4-week treatment period
  Other Names: Coreg
  Arms: Carvedilol 2.5 mg
Drug: Placebo capsule — Participants will receive a matching oral dose of placebo capsule twice daily during the 4-week treatment period
  Arms: Placebo capsule

SUMMARY:
Type 1 diabetes mellitus (T1DM) can lead to cardiovascular, renal and neurological complications if left poorly-controlled over prolonged periods of time. However, lowering glycemic goals for diabetic patients increases their risk for hypoglycemia exposure. Hypoglycemia is associated with symptoms such as heart palpitations, fatigue, shakiness, anxiety, confusion, and blurred vision. Recurrent hypoglycemia leads to impairment of the body's autonomic and symptomatic responses to this condition, and can result in loss of awareness in the patient of the hypoglycemic state. Repeated incidences of hypoglycemia from loss of this awareness can result in even more hypoglycemic episodes and more severe outcomes, such as loss of consciousness, accidents, hospitalization and even death if left untreated.

The aim of this study is to investigate whether adrenergic blockade through the use of low-dose carvedilol treatment can improve hypoglycemia awareness and the counterregulatory hormone responses to hypoglycemia in T1DM patients with impaired awareness of hypoglycemia.

DETAILED DESCRIPTION:
Hypoglycemia elicits a multifaceted hormonal response that helps restore glycemic levels to normal. As blood glucose levels start to fall, insulin secretion ceases. At the top of this hierarchy of counterregulatory responses are glucagon and epinephrine which are the two principal hormones that act rapidly to increase glucose production and inhibit glucose utilization to raise plasma glucose levels back to normal. In cases of prolonged and/or more severe hypoglycemia, growth hormone and cortisol are mobilized to stimulate the synthesis of gluconeogenic enzymes and inhibit glucose utilization. In non-diabetic individuals, glucagon and epinephrine are usually very effective and the latter responses are rarely required in the acute situation. In contrast, impaired glucose counterregulation presents itself in longstanding diabetes and with antecedent hypoglycemia. Within the first five years after the onset of T1DM, the primary defense against hypoglycemia, the release of glucagon, either becomes significantly attenuated or is completely absent in diabetic patients and this impairment appears to be specific for the stimulus of hypoglycemia. Hence, patients with diabetes primarily depend on the release of epinephrine as their main defense against hypoglycemia. Unfortunately, with longer duration of diabetes and especially with poor glycemic control, epinephrine secretion is also compromised, making these patients even more vulnerable to the threat of hypoglycemia. In patients with diabetes, hypoglycemia arises from the interplay of a relative excess of exogenous insulin and defective glucose counterregulation and it remains a limiting factor in attaining proper glycemic management. Both the Diabetes Control and Complications Trial (DCCT) conducted in Type 1 patients and the United Kingdom Prospective Diabetes Study (UKPDS) conducted in Type 2 patients, have established the importance of maintaining good glucose control over a lifetime of diabetes to avoid cardiovascular, renal and neurological complications. However, lowering glycemic goals for diabetic patients increases their risk for hypoglycemia exposure. According to the DCCT, T1DM patients put on intensive insulin therapy, though having improved outcomes for diabetic complications, are at a 3-fold higher risk of experiencing severe hypoglycemia compared to those on conventional insulin therapy. Moreover, recent antecedent hypoglycemia reduces autonomic (epinephrine) and symptomatic (which normally prompts behavioral defenses such as eating) responses to subsequent bouts of hypoglycemia. Thus begins the vicious cycle of recurrent hypoglycemia (RH) where hypoglycemia leads to further impairment of counterregulatory responses which tin turn, begets more hypoglycemia and so forth. Because of the imperfections of current insulin therapies, those patients attempting to achieve glycemic control suffer an untold number of asymptomatic hypoglycemic episodes. Current estimates of symptomatic hypoglycemic episodes range form 2-3 incidences per week on average and severe, debilitating episodes occur one or twice each year. Therefore, developing therapies to prevent or eliminate hypoglycemia is of great importance.

Sensors that detect changes in blood glucose levels and initiate glucose counterregulatory responses have been identified in both the periphery and within the brain. These sensors have been localized to the hepatic portal vein, the carotid body and the brain. In the brain, the dominant sensors are located in the hypothalamus. While peripheral glucose sensors may play a role in mediating the immediate counterregulatory responses to hypoglycemia, it is thought that glucosensors located within the brain may have a redundant regulatory and/or modulatory role in regulating glucose counterregulatory responses. It is well established that brain glucose sensors are crucial for detecting falling blood glucose levels and for initiating counterregulatory responses. These sensors are located in the hindbrain, the lateral hypothalamus, the paraventricular nucleus, the dorsal hypothalamus and the ventromedial hypothalamus (VMH). The neurons within the VMH contain much of the same glucose sensing machinery as the pancreatic β-cells. To date, two main types of glucose sensing neurons have been identified in the brain - those that increase their firing rate in response to increases in glucose levels, the "glucose-excited" (GE) neurons and those that decrease their firing rate in response to increases in glucose levels, the "glucose-inhibited" (GI) neurons. The mechanism by which GE neurons sense changes in blood glucose concentrations is believed to be similar to that used by pancreatic β-cells whereas GI neurons respond to decreases in ambient glucose levels through activation of the metabolic fuel sensor, AMP kinase (AMPK), and closure of chloride channels that result in increased activity of GI neurons. Although many of these sensing components have been identified, it is still not entirely clear how glucose sensing neurons regulate counterregulatory hormone release. It has been proposed that alterations in the firing rates of VMH glucose sensing neurons in response to glucose or fuel deficits can inhibit (as is the case for GE neurons) or stimulate (as is the case for GI neurons) the exocytosis of vesicles containing neurotransmitters that can modulate the counterregulatory hormone response.

The inhibitory neurotransmitter, GABA, and the stimulatory neurotransmitters, glutamate and norepinephrine (NE), act within the VMH to suppress or stimulate the counterregulatory responses to hypoglycemia, respectively. In response to an initial bout of hypoglycemia, VMH GABA levels decrease while glutamate and NE levels increase, allowing for activation of the counterregulatory hormone responses. While these studies underscore the importance of VMH neurotransmitter signaling in regulating glucose homeostatic mechanisms, to date, the mechanisms that lead to their dysregulation in models of counterregulatory failure are not entirely clear. Recent evidence suggests that lactate, which serves as an alternate fuel substrate in the brain, plays an important role in precipitating the defects noted above. Lactate produced from neighboring astrocytes can supplement higher energy requirements during periods of increased neuronal activity or when glucose supply is limited. If this is the case, then lactate can be used in place of glucose as a fuel for VMH glucose sensing neurons, preventing them from detecting a fall in glucose levels, causing (inhibitory) GABA tone to be enhanced and (stimulatory) glutamate output to be reduced. Together, these actions ultimately suppress the release of counterregulatory hormones. In recent years, it has been shown that lactate levels are sensed by the brain and more specifically, can act in the hypothalamus to regulate glucose homeostasis, appetite and body weight. Lactate prevents the activation of hypothalamic neurons during glucose deprivation and more pertinent to this application, attenuates glucose counterregulatory responses to hypoglycemia when locally administered into the VMH. Data from the investigator's research group revealed VMH extracellular lactate concentrations are elevated in RH and diabetic animals and in particular, these conditions also increase expression of the lactate transporter in the VMH. When VMH lactate uptake is pharmacologically inhibited, neurotransmitter and counterregulatory responses improve in both RH and diabetic animals, suggesting lactate plays an important role in dysregulating neurotransmitter systems in the VMH, which in turn, impairs counterregulatory responses. Preliminary data suggests that therapeutic strategies that can reduce brain lactate levels, may help restore hypothalamic glucose sensing mechanisms and the counterregulatory response to hypoglycemia. Hence, identifying the mechanisms that increase VMH lactate levels may lead to suitable therapeutic strategies to prevent hypoglycemia.

Norepinephrine can enhance lactate production from astrocytes and it can also increase the uptake of lactate into neurons through the activation of β2-adrenergic receptors (β2AR), potentially helping to coordinate both the supply and uptake of lactate into neurons. Normally, in response to an acute bout of hypoglycemia, VMH NE levels rise and act through β2ARs to enhance the sympathoadrenal response. Although activation of VMH β2ARs augments the counterregulatory response during acute bouts of hypoglycemia, less is known about the effects of RH on this neurotransmitter system. It has been reported that VMH NE levels are not altered by successive bouts of hypoglycemia, suggesting activation of the VMH NE system is not dampened by RH and that its suppressive effects on counterregulatory hormone release may lie downstream of NE release. In support of this finding, adrenergic blockade during antecedent bouts of hypoglycemia was shown to prevent counterregulatory failure in healthy human subjects. Therefore, while acute activation of VMH adrenergic receptors may be beneficial in its capacity to enhance the counterregulatory response, repeated activation of this neurotransmitter system may contribute to counterregulatory failure, but the mechanisms by which this occurs have not been fully identified.

To evaluate whether repeated activation of the VMH NE system contributes to counterregulatory failure, NE was microinjected into the VMH of non-diabetic, hypoglycemia-naive rats for 3 hours/day for 3 consecutive days before subjecting the animals to a hypoglycemic glucose clamp on day 4. Repeated activation of the VMH NE system in the absence of hypoglycemia, increased VMH lactate levels and more importantly, blunted the counterregulatory hormone responses to hypoglycemia. This phenomenon was recapitulated with microinjection of salbutamol, a short-acting β2AR agonist, into the VMH using the same protocol as for NE, suggesting the suppressive effects of NE are mediated through VMH β2ARs. In a subgroup of animals treated with NE, uptake of lactate into neurons was blocked immediately prior to the hypoglycemic clamp. In this group, the suppressive effects of NE treatment on glucose counterregulation were completely abolished. Hence, preliminary data suggests that repeated activation of the VMH NE system plays a role in the development of counterregulatory failure, in part by enhancing central lactate production and therefore, the use of β-adrenergic blockers may be a promising treatment to preserve the responses to hypoglycemia. Preliminary data show that RH rats treated with low doses of the non-specific β-blocker, carvedilol, during the induction of RH, required less exogenous glucose during the hypoglycemic clamp compared to RH animals treated with vehicle. More importantly, reductions in VMH lactate levels and significant improvements in the counterregulatory hormone responses to hypoglycemia in the carvedilol-treated RH animals were observed.

Carvedilol is a third generation non-selective, vasodilating β-blocker, which is FDA-approved for the treatment of congestive heart failure and hypertension. Carvedilol mainly blocks β2- and β1-adrenergic receptors and some α1-adrenergic receptors. Due to its lipophilic nature, carvedilol readily crosses the blood-brain barrier. As the brain is the primary target, this beneficial pharmacokinetic property of carvedilol improves central nervous system bioavailability, allowing lower doses to be used to deliver treatment to the brain. With lower doses, the potential for side effects stemming from unnecessary exposure of peripheral tissues to high levels of β-adrenergic blockade can be reduced. This study is designed to evaluate the effectiveness of low-dose carvedilol treatment for 4 weeks as a treatment for restoring the counterregulatory hormone responses to hypoglycemia and improve hypoglycemia awareness in T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* History of Type 1 diabetes mellitus for more than 5 years
* Age > 18 years
* Presence of impaired hypoglycemia awareness/unawareness
* Intensive insulin treatment as defined by multiple daily insulin injections (3 or more) or insulin pump therapy
* Negative pregnancy test
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Major medical disorders (including liver disease, cardiovascular disease, kidney disease, chronic obstructive pulmonary disease, asthma, active malignancy or HIV)
* Overt diabetes complications (neuropathy, nephropathy, retinopathy)
* Presence of anemia
* Current or recent use of beta-blocker therapy
* Use of diuretics
* Allergies or contraindications to beta-blockers or heparin
* Use of benzodiazepines
* Alcohol, drug or medication abuse
* Frequent use of acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen Chan, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Started | 0 | 0 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study was terminated early and there were 0 participants enrolled into the Carvedilol 3.125 mg arm and 0 participants enrolled into the Carvedilol 2.5 mg arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule | Total
Number analyzed (Participants) | 0 | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 1 | 1
  >=65 years |  |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 1 | 1
  Male |  |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 0 | 0
  Not Hispanic or Latino |  |  | 1 | 1
  Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 0 | 0
  White |  |  | 1 | 1
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hypoglycemia Symptom Score
Description: Participants will complete the Edinburgh Hypoglycemia Symptom questionnaire at baseline and after the 4-week treatment period. The average change in hypoglycemia symptom score will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: Study terminated due to low enrollment. Subject did not complete the study and data were not collected to enable results reporting.
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Blood Glucagon
Description: Blood samples will be drawn from study participants at baseline and after the 4-week treatment period during the clamp procedure. The average change in blood glucagon level will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Blood Epinephrine
Description: Blood samples will be drawn from study participants at baseline and after the 4-week treatment period during the clamp procedure. The average change in blood epinephrine level will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Blood Norepinephrine
Description: Blood samples will be drawn from study participants at baseline and after the 4-week treatment period during the clamp procedure. The average change in blood norepinephrine level will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Blood Cortisol
Description: Blood samples will be drawn from study participants at baseline and after the 4-week treatment period during the clamp procedure. The average change in blood cortisol level will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Blood Growth Hormone
Description: Blood samples will be drawn from study participants at baseline and after the 4-week treatment period during the clamp procedure. The average change in blood growth hormone level will be compared between the carvedilol and placebo groups.
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Frequency of CGM-Determined Hypoglycemic Episodes
Description: The number of hypoglycemic episodes as determined by CGM will be determined during the 4-week treatment period and compared to the 1-week pre-study baseline period.
Time Frame: 5 Weeks
Population: as for outcome 1
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 Weeks
Description: Study was terminated early and there were 0 participants enrolled into the Carvedilol 3.125 mg arm and 0 participants enrolled into the Carvedilol 2.5 mg arm.
Arm/Group | Carvedilol 3.125 mg | Carvedilol 2.5 mg | Placebo Capsule
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03538015/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03538015/ICF_001.pdf